CLINICAL TRIAL: NCT01601418
Title: Double-blind, Placebo-controlled, Single-dose, 5-way Crossover Study of the Effect of YF476 (1, 5, 25 & 100 mg) on Pentagastrin-induced Gastric Acid Output in Healthy Volunteers
Brief Title: Effect of Single Doses of YF476 on Stomach Acidity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Trio Medicines Ltd. (Industry)
Collaborators: James Black Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 01-022
Record Dates: First submitted 2012-05-15; First posted 2012-05-18 (Estimated); Last update posted 2012-05-18 (Estimated); Status verified 2012-05

CONDITIONS: Hypergastrinaemia
Keywords: YF476; gastrin receptor antagonist; pentagastrin; gastric acid; healthy subjects
MeSH Terms: interventions — YF 476

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: YF476 — Each subject took one capsule of YF476 (1, 5, 25 or 100 mg) or placebo on five separate occasions. Each capsule was taken with water 150 mL.
Drug: Placebo — Each subject took one capsule of YF476 (1, 5, 25 or 100 mg) or placebo on five separate occasions. Each capsule was taken with water 150 mL.

SUMMARY:
The objective of the study was to assess the effect of a range of single oral doses of YF476 on pentagastrin-induced gastric acid output in healthy volunteers

DETAILED DESCRIPTION:
The rationale for the study was as follows.

On the basis of the pre-clinical studies, the original target disease for YF476 was gastro-oesophageal reflux disease (GORD), not only because of the excellent anti-secretory activity of YF476 but also because of its potential for increasing gastric emptying. But loss of the anti-secretory effect of YF476 in healthy subjects after repeated dosing excludes its use as an anti-secretory agent in patients with GORD. However, there is some evidence from within our repeated-dose studies in healthy subjects that gastrin receptors are blocked despite loss of the anti-secretory activity of YF476. Further evidence that repeated doses of YF476 cause sustained blockade of gastrin receptors comes from several types of study in animals. First, in the 13-week toxicology studies, all dose levels of YF476 reduced the ECL population, unlike other anti-secretory agents, histamine H2-antagonists and proton-pump inhibitors, which increase the ECL population. Second, YF476 at doses of 0.1 and 1.0 mg/kg subcutaneously twice daily for 14 days in rats abolished the increase in gastric output induced by pentagastrin on Days 1, 7 and 14.

This protocol describes a study in healthy subjects using inhibition of pentagastrin-induced gastric acid output as a surrogate marker of efficacy of YF476. Pentagastrin has been used for many years to test gastric function in healthy subjects and patients. Intravenous infusion of 0.6 micrograms/kg/hour is a submaximal and well-tolerated dose.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female volunteers.
* Aged 18-45 years.
* A body mass index (Quetelet index) in the range 18.0-30.9.
* Women at risk of pregnancy must use a reliable method of contraception.
* No clinically relevant abnormal findings in the clinical history or physical examination at the screening assessment which could interfere with the objectives of the study or make the volunteer's participation hazardous.
* No clinically relevant abnormal laboratory values at the screening evaluation, including a normal ECG.
* Sufficient intelligence to understand the nature of the study and any hazards of participating in it. Ability to communicate satisfactorily with the investigator and to participate in, and comply with the requirements of, the entire study.
* Willingness to give written consent to participate after reading the Consent Form, and after having the opportunity to discuss the study with an investigator or his deputy.

Exclusion Criteria:

* Women who are pregnant or lactating.
* Clinically relevant abnormal history, physical findings, ECG, or laboratory values at the pre-study screening assessment that could interfere with the objectives of the study or the safety of the volunteer.
* Presence of acute or chronic illness or history of chronic illness sufficient to invalidate the volunteer's participation in the study or make it unnecessarily hazardous.
* Positive test for Helicobacter pylori.
* Impaired endocrine, thyroid, hepatic, respiratory or renal function, diabetes mellitus, coronary heart disease, or history of any psychotic mental illness.
* Presence or history of severe adverse reaction to any drug or a history of severe allergic disease.
* Use of a prescription medicine (except oral contraceptives in females) during the 30 days before the study or use of an over-the-counter medication, with the exception of paracetamol, during the 7 days before the study.
* Participation in other clinical studies of a new chemical entity or a prescription medicine within the previous 3 months.
* Smokers.
* Presence or history of drug or alcohol abuse, or intake of more than 28 units of alcohol weekly (for men) or 21 units of alcohol weekly (for women).
* Blood pressure and heart rate in seated position at the screening examination outside the ranges 90-160 mm Hg systolic, 40-95 mm Hg diastolic; heart rate 40_100 beats/min.
* Possibility that the volunteer will not cooperate with the requirements of the protocol.
* Evidence of drug abuse on urine testing.
* Positive test for hepatitis B, hepatitis C, HIV1 or HIV2.
* Loss of more than 400 mL blood during the 3 months before the study, e.g. as a blood donor.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2001-10; Primary Completion 2002-01 (Actual); Study Completion 2002-01 (Actual)

PRIMARY OUTCOMES:
Safety of YF476 | 12 weeks
  Assessed by medical examinations, ECG, safety tests of blood and urine
Tolerability of YF476 | 12 weeks
  Assessed by adverse events
Efficacy of YF476 | 12 weeks
  Comparison of YF476 doses and placebo with respect to:
  1. area under the total H+ secretion, i.e. [H+] x volume-time curve (corrected for basal secretion)
  2. peak total H+ secretion, i.e. [H+] x volume-secretory rate (corrected for basal secretory rate)

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm Boyce, Study Director — Trio Medicines Limited
Locations (1):
- Hammersmith Medicines Research, London, United Kingdom